CLINICAL TRIAL: NCT02918695
Title: Comparison of Different Geriatric Screening Methods in Newly Diagnosed Multiple Myeloma Patients, and Assessment of Therapeutic Efficacy and Toxicity in Fit and Frail Patients. A Multicenter Observational Belgian Study.
Brief Title: Comparison of Geriatric Screening Methods in Newly Diagnosed Multiple Myeloma Patients
Acronym: COMPASS
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: NA-NI-MM-PI-006760
Record Dates: First submitted 2016-09-13; First posted 2016-09-29 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma; Hematologic Diseases
Keywords: Geriatric assessment; Fit and frail elderly; Geriatric oncology
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to compare clinical judgment and comprehensive geriatric assessment as screening tools for optimization of treatment for newly diagnosed elderly multiple myeloma patients.

DETAILED DESCRIPTION:
Given the growing elderly multiple myeloma population, the increase in therapeutic possibilities and the importance of geriatric screening, this study wants:

* to compare clinical judgment with standardized geriatric screening approaches (G8, CGA and IMWG score) in newly diagnosed elderly myeloma patients and to evaluate their influence on the detection of geriatric problems and on the choice of the anti-myeloma treatment
* to evaluate how geriatric scoring and the subsequent treatment choice influences the therapeutic efficacy and toxicities

Geriatric scoring will be performed in 3 different ways:

* by clinical judgment performed by the treating physician
* by validated scoring systems independently performed by a trained nurse/ health care worker. Initial scoring will be done by the G8 score. If an abnormal G8 score is present (<= 14), CGA will be performed.
* based on the CGA parameters, the Palumbo/IMWG geriatric score will be calculated

Results obtained by physician-based assessment and by geriatric assessment will be compared before treatment initiation. If, and to what extent the knowledge of the GA influences the therapeutic decision of the treating physician will be registered. In addition, we will register which geriatric problems diagnosed by the CGA assessment were already known or unknown by the treating physician. After three months of treatment and at the time of disease progression, geriatric assessment will be repeated in order to judge the evolution (disappearance, improvement, worsening) of the scored parameters, or the emergence of new geriatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed multiple myeloma
* age => 70 years
* no previous anti-myeloma treatment except for local radiotherapy or short course (max 4 days) of high-dose dexamethasone
* signed informed consent
* patients included in an interventional therapeutic trial are eligible

Exclusion Criteria:

* previous systemic anti-myeloma treatment
* severe mental or cognitive disorder precluding geriatric assessment
* patient refusal to sign informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 200 newly diagnosed elderly Multiple Myeloma patients
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the geriatric categorization (fit versus frail) by standard clinical assessment versus by geriatric scoring. | At baseline
  Comparison of geriatric categorization by standard clinical assessment (fit versus frail ) versus by geriatric scoring ( G8 score, CGA (Comprehensive Geriatric Assessment) and IMWG score will result in fit or frail) will be presented in proportion of agreement (accuracy, specificity, sensitivity, positive predictive value, negative predictive value).

SECONDARY OUTCOMES:
Comparison of the geriatric categorization (fit versus frail) by CGA versus by IMWG scoring | At baseline
  The results will be presented in terms of accuracy, specificity, sensitivity, positive predictive value, negative predictive value.
Change in geriatric categorization (fit versus frail) by CGA from baseline to 3 months of anti-myeloma therapy. | after 3 months of anti-myeloma treatment
Change in geriatric categorization (fit versus frail) by CGA from baseline to time of first relapse of multiple myeloma | At first relapse of multiple myeloma, defined according to IMWG criteria (ref. Durie et al. Leukemia 2006)
Description of geriatric problems detected by CGA ( unknown items assessed by validated CGA scoring tool)(ref. Kenis et al. An of Onc 2013;24:1306) | At baseline
Response rate | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.
Progression free survival | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.
Overall survival | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.
Treatment-related deaths | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.
Grade 3 and 4 non-hematological and grade 4 hematological adverse events (according to CTCAE 4.0) | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.
Treatment discontinuation | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.
Dose reductions of anti-myeloma treatment | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.
Description of the causes for dose-reduction and/or treatment discontinuation | Up to 1 year after signing the informed consent, or until disease progression, until anti-myeloma treatment discontinuation, until withdrawal of informed consent, until death or loss to follow-up, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delforge, MD PhD, Principal Investigator — UZ Leuven Gasthuisberg
Locations (20):
- Belgium (20):
  - ZNA Antwerpen, Antwerp
  - Centre Hospitalier EpiCURA, Baudour
  - Imelda Ziekenhuis, Bonheiden
  - AZ Klina, Brasschaat
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - GHdC Charlerloi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - UZ Gent, Ghent
  - Hôpital de Jolimont, Haine-Saint-Paul
  - Jan Yperman Ziekenhuis, Ieper
  - AZ Groeninge, Kortrijk
  - CHU Tivoli, La Louvière
  - UZ Leuven Gasthuisberg, Leuven
  - Heilig-Hartziekenhuis Lier, Lier
  - CHU de Liège, Liège
  - AZ Nikolaas, Sint-Niklaas
  - CHU Dinant-Mont-Godinne, Yvoir